CLINICAL TRIAL: NCT00897091
Title: Molecular Predictors of Outcome on CAF Plus Tamoxifen Versus Tamoxifen Alone in Postmenopausal Women With Node Positive, Receptor Positive Breast Cancer [NCI Correlative Science Reference No. # 8814A-ICSC]
Brief Title: S8814A Biomarkers in Predicting Outcome in Postmenopausal Women With Hormone Receptor-Positive, Node-Positive Breast Cancer Treated With Tamoxifen With or Without Cyclophosphamide, Doxorubicin, and Fluorouracil
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000528264; S8814A-ICSC (Other: SWOG); GHI-01-024 (Other: Genomic Health); U10CA032102 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Comparative Genomic Hybridization; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: comparative genomic hybridization
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers in predicting outcome in postmenopausal women with hormone receptor-positive, node-positive breast cancer treated with tamoxifen with or without cyclophosphamide, doxorubicin, and fluorouracil.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the value of the Oncotype DX Recurrence Score for prediction of treatment benefit of cyclophosphamide, doxorubicin hydrochloride, and fluorouracil (CAF) chemotherapy, in terms of disease-free survival (DFS) and overall survival (OS), in postmenopausal patients with estrogen and/or progesterone receptor-positive, node-positive breast cancer treated on clinical trial SWOG-8814.
* Determine the overall prognostic value of the Oncotype DX Recurrence Score, in terms of DFS and OS, in patients treated with tamoxifen citrate alone or CAF with concurrent or sequential tamoxifen citrate.

Secondary

* Determine the optimal cut point (i.e., low, intermediate, and high recurrence risk) for the Recurrence Score in these patients.
* Determine the relationship between expression of any one of the 21 genes on the Oncotype DX gene panel with DFS and OS.
* Determine whether the expression of any of these genes are associated with CAF treatment benefit.
* Determine the relationship between the Oncotype DX Recurrence Score and DFS and OS in multivariate models, including number of positive nodes, tumor size, tumor grade, estrogen receptor, progesterone receptor, and HER2 and p53 status.
* Determine the relationship between quantitative reverse-transcriptase-polymerase chain reaction expression of up to 800 additional genes and prognosis and/or prediction of CAF benefit.

OUTLINE: This is a multicenter study.

Fixed paraffin-embedded breast tumor tissue samples (obtained from the SWOG Central Tumor Repository at the University of Colorado) are analyzed by the Oncotype DX panel containing the following 21 genes: BAG1, Bc12, CCNB1, CD68, SCUBE2, CTSL2, Esrt1, GRB7, GSTM1, HER2, Ki-67, MYBL2, PR, STK15, STMY3, SURV, B-actin, GAPDH, GUS, RPLPO, and TFRC. The Oncotype DX Recurrence Score is calculated for each patient. Analyses are performed to determine the relationship between the Recurrence Score and gene expression and prognosis/prediction of therapy (tamoxifen citrate alone or cyclophosphamide, doxorubicin hydrochloride, and fluorouracil with concurrent or sequential tamoxifen citrate) benefit as well as to determine the relationship between clinical and demographic covariates and disease-free and overall survival.

Samples are also analyzed by reverse-transcriptase-polymerase chain reaction for exploratory analysis of up to 800 additional genes that may be prognostic and/or predict the likelihood of therapy benefit.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Node-positive disease (pT1-3a, pN1-2 [clinical N0-1], M0)
* Previously enrolled in SWOG-8814, a treatment clinical trial, and in SWOG-9445, a companion tissue banking study
* Tumor block or unstained sections available from initial diagnosis in the SWOG archive

  * Sufficient tumor in block or unstained sections
  * Patients for whom only unstained slides are available must have acceptable reverse-transcriptase-polymerase chain reaction (RT-PCR) profiles
* Sufficient RNA (≥ 300 ng) for RT-PCR analysis with the Oncotype DX 21 gene assay
* Average normalized cycle threshold for the 5 reference genes ≤ 35
* Follow-up data from the SWOG-8814 clinical trial obtained from the patient
* Hormone receptor status:

  * Estrogen and/or progesterone receptor positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consenting to banking in S8814
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival
Overall survival

SECONDARY OUTCOMES:
Distant disease-free recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Kathy S. Albain, MD, Study Chair — Loyola University
Locations (1):
- Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois, United States